CLINICAL TRIAL: NCT02993562
Title: Levothyroxine Substitution Therapy in Hypothyroid Patients - Impact on Appetite and Food Intake
Brief Title: Hypothyroidism, Metabolism and Food Intake
Acronym: Hypomafia
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Center for Diabetes Research, Herlev and Gentofte Hospital. (Unknown)
Responsible Party: Principal Investigator, Bjarke Borregaard Medici, Principial Investigator, Herlev Hospital
Other Study IDs: Herlev-Gentofte Hypomafia
Record Dates: First submitted 2016-10-20; First posted 2016-12-15 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Hypothyroidism
Keywords: Food intake; Resting Energy Expenditure; Gall Bladder emptying; Insulin response; Body Composition
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypothyroid patients: Hypothyroid patients treated with Levothyroxine as part of normal treatment.
  Interventions: Drug: Levothyroxine
- Healthy volunteers: Matched on age and BMI. 18 Persons.

INTERVENTIONS:
Drug: Levothyroxine — Normal treatment with levothyroxine.
  Other Names: Eltroxin/Euthyrox
  Groups: Hypothyroid patients

SUMMARY:
This project has the following primary aims:

To measure changes in appetite and food intake in newly diagnosed hypothyroid patients during the first six months after starting levothyroxine (L-T4) substitution therapy

Secondary aims are:

To delineate the effect of L-T4 substitution therapy on thyroid status, body weight, body mass index (BMI), body composition, physical activity, glycaemic control, postprandial gut and pancreatic hormone responses, gastric and gall bladder emptying, resting energy expenditure (REE), quality of life (QOL) and cognitive function

DETAILED DESCRIPTION:
18 newly diagnosed hypothyroid female patients and 18 healthy controls age between 20 and 75 years will be recruited from the out-patients clinic in Herlev and Gentofte Hospital and the general practitioners before start of substitution therapy.

The study is devided in to three identical experimental days of approx. 6 hours. First experimental day placed before T4 treatment is initiated. Second day as soon as Thyroid Stimulating Hormone (TSH) is below 4 milli unit pr liter (mU/l). The Third experimental day after 6 months of T4 therapy.

For 5-7 days before each experimental day, the participants' physical activity energy expenditure (PAEE) will be monitored by an Actiheart® pedometer attached to the skin of the chest.

The last two days before each experimental day, the participants will follow a standardised diet following World Health Organization guidelines on energy requirements and nutrient composition according to gender, age and body weight Shortly after diagnosis patients will undergo a test panel at the first experimental day, where patients arrives fasting.

Visual analog score on satiety and thirst will be filled out continuously. REE will be measured by a CCM-express calorimeter,

* Dual Energy X-ray absorptiometry (DEXA)-scan
* Blood samples will be taken continuously during the experimental day. Gall bladder size will be examined at 6 times during the experimental day using ultra sound.

At the end of the day, patients´ satiety will be examined with an ad libitum meal.

Blood will be analysed for Gastric inhibitory polypeptide (GIP), Glucagon-like Peptide 1 (GLP-1), Glucagon-like Peptide 2 (GLP-2), glucagon, peptide tyrosine tyrosine (PYY), Gastrin, Cholesystokinin (CCK), Insulin, C-peptide, Blood sugar, Cholesterol, Free fatty acids and paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* TSH > 10
* Female

Exclusion Criteria:

* Competing serious disease
* Male
* Not able to understand written and spoken danish
* Pregnancy
* Thyroidectomized patients
* Amiodarone treatment.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 Hypothyroid female patients with a TSH > 10 without Levothyroxine treatment.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-08; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in food intake at ad libitum meal | 6 months
  Changes in food intake at ad libitum meal measured at each experimental day
Satiety | 6 months
  Satiety measured on a visual analog score 13 times during each experimental day.

SECONDARY OUTCOMES:
Changes in lean mass assessed through lean mass | 6 months
  Changes in lean mass assessed through lean mass with DEXA-scan
Changes in fat mass assessed through lean mass with DEXA-scan | 6 months
  Changes in lean mass assessed through lean mass with DEXA-scan
Changes in gall bladder emptying | 6 months
  Changes in gall bladder emptying evaluated with ultrasound 6 times each experimental day before and after meal.
Changes in resting energy expenditure | 6 months
  Changes in resting energy expenditure measured 3 times each experimental day using Indirect Calorimetry.
Changes in blood sugar response to standardized meal. | 6 Months
  changes in blood sugar response to standardized meal measured before and after meal at each experimental day.
Changes in stomach emptying | 6 months
  Evaluated with continously measuring serum paracetamol after standardized meal containing 1,5 g paracetamol.
Changes in GIP hormones | 6 months
  Continously measuring of a range of hormones during each experimental day: GIP
Changes in GLP-1 hormones | 6 months
  Continously measuring of GLP-1 hormones during each experimental day
Changes in GLP-2 hormones | 6 Months
  Continuously measuring of GLP-2 hormones during each experimental day
Changes in PYY hormones | 6 Months
  Continuously measuring of PYY hormones during each experimental day
Changes in CCK hormones | 6 Months
  Continuously measuring of CCK hormones during each experimental day
Changes in Gastrin hormones | 6 Months
  Continuously measuring of Gastrin during each experimental day
Changes in Insulin hormones | 6 Months
  Continuously measuring of Insulin during each experimental day
Changes in Glucagon | 6 Months
  Continuously measuring of Glucagon during each experimental day
Changes in C-peptide | 6 Months
  Continuously measuring of C-peptide during each experimental day
Changes in Free-Fatty acids | 6 Months
  Continuously measuring of Free Fatty acids during each experimental day

CONTACTS AND LOCATIONS:
Overall Officials: Bjarke B Medici, MD, Principal Investigator — Department of Internal Medicine, Herlev and Gentofte hospitals.
Locations (1):
- Center for Diabetes Research, Herlev and Gentofte Hospitals, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No